CLINICAL TRIAL: NCT07082764
Title: A Phase 2a Safety and Efficacy Study of TAR-0520 Gel in Prevention of Taxane-induced Peripheral Neuropathy
Brief Title: Safety and Efficacy Study of TAR-0520 Gel in Prevention of Taxane-induced Peripheral Neuropathy
Acronym: TARIAN 014
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tarian Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TARIAN 014; 2025-521674-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-03; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy Induced Peripheral Neuropathy
Keywords: taxane-induced peripheral neuropathy; taxane-induced nail toxicities

STUDY DESIGN:
Intervention Model Description: intra-individual comparaison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intra-individual active comparator vs no intervention (Experimental): Tar-0520 gel will be applied to one hand and to homolateral foot ,other hand and foot will be not treated and will serve as control
  Interventions: Drug: Brimonidine gel; Other: No intervantion

INTERVENTIONS:
Drug: Brimonidine gel — TAR-0520 gel
Other: No intervantion — No treatment

SUMMARY:
Taxane -induced peripheral neuropthy (TIPN) and nail toxicites are frequent side effects of taxane therapy in breast cancer patients.. TIPN involves the hands and the feet ,its symptoms comprise numbness,tingling,altered touch sensation, impaired vibration, parasthesia and dysesthesias induced by touch, warm or cool temperatures.

This study investigate the preventive effect of TAR-0520 gel on TIPN and on nail toxicity.

Breast cancer patients under taxanes therapy will apply TAR-0520 Gel to one hand and the homolateral foot including fingers and toes. Other hand and foot will be untreated and will serve as control.

Patients will be followed during the 12 cycles of taxane therapy. Evaluations of TIPN will include clinical assessments by the oncologist, examination by a neurologist, patient questionnaires administered by a nurse and objective neurophysiological measures conducted by trained personnel. Evaluation of taxane nail toxicity will include a clinical grading by a nurse and a patient questionnaire.

DETAILED DESCRIPTION:
This is a Phase 2a, open label, intra-individual study with approximately 30 patients included.

Principal objective of the study is to confirm the local and systemic safety of TAR-0520 Gel applied twice daily to one hand and one foot, in breast cancer patients treated with taxanes.

Secondary objectives of the study are:

* To explore the preventative effect of TAR-0520 Gel on taxane-induced TIPN,
* To explore the preventative effect of TAR-0520 Gel on taxane-induced onycholysis and other nail changes.

Each patient will receive the active drug candidate TAR-0520 gel for 3 days at each taxane cycle (usually 12 cycles with an infusion every week). During these 3 days, TAR-0520 gel will be applied to one hand and one foot, twice daily, starting the day of taxane infusion and continuing the next two days (thus covering the period when Paclitaxel will be circulating: elimination half-life of the drug is approximately 24 hours).

TAR-0520 gel will be applied by the patients themselves using their dominant hand wearing a glove, patients will apply TAR-0520 gel to the contro-lateral hand and foot. Test product is to be applied to both palmo-plantar and dorsal areas of hand and foot including fingers/toes and the skin surrounding nails. No product is to be applied to the hand and foot on the other side (dominant hand side).

Patients will be included one week before the taxane treatment initiation and followed during the 12 taxane cycles as well as 12 weeks later (follow-up visit). Evaluations of TIPN will include clinical assessments by the oncologist, examination by a neurologist, patient questionnaire administered by a nurse and objective neurophysiological measures conducted by trained personnel. Evaluation of nail toxicities will include clinical grading by a nurse and a patient questionnaire.

The study will include 17 visits: a Screening visit, 15 evaluations visits and a follow-up visit (Final assessment) that will occur approximately 12 weeks after the last taxane infusion.

Evaluations visits will be conducted one week before the first taxane infusion, the days of taxane infusions, between the 6th and the 7th cycle of taxane infusion, one week after the last taxane infusion and at a follow-up visit, 3 months after the last taxane infusion. This design will allow to assess TIPN progression during treatment as well as persistent TIPN following treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, who is at least 18 years of age or older
* Patients with clinical diagnosis of breast cancer
* Patients planned to be treated with paclitaxel or docetaxel
* Patients who can understand and sign the Informed Consent Form
* Patients who can apply the study gel by himself /herself or has a giver that can apply the product.
* Female patients of childbearing potential who agree to use a highly effective method of contraception throughout the study

Exclusion Criteria:

* Patient already treated with taxanes or other chemotherapies known to induce neuropathies
* Patient with previously diagnosed peripheral neuropathy
* Patient with concomitant therapies known to induce neuropathies
* Patient treated for neuropathic pain
* Patient with comorbid factors known to induce neuropathies (such as Diabetes, Alcoholism, HIV, Peripheral vascular disease, Vitamin B deficiencies)
* Patient currently receiving monoamine oxidase (MAO) inhibitors therapy or patients on antidepressants which affect noradrenergic transmission e.g. tricyclic antidepressants and mianserin (as mentioned in the current topical brimonidine labeling of approved products).
* Patient who will not be able to follow the protocol for physical or psychological reasons
* Patient with history of skin disorders, significant skin disease, irritated skin or open wounds within the same body areas planned for the IMP application.
* Known or suspected allergies or sensitivities to any components of any of the study drugs (see Investigator's Brochure/Product label)
* Female who is pregnant or lactating
* Female who intends to conceive a child during the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Number of treatment related local adverse events | From Baseline up to the end of 12 taxane perfusions
  Treatement related local adverse events inluding erythema, oedema, pruritus

SECONDARY OUTCOMES:
CTCAE grade of peripheral neuropathy | From Baseline up to the end of 12 taxane perfusions
  CTCAE V5.0 Nervous system disorders grading ( Grade 0-5, 0-asymptomatic, 5- death)
Instrumental objective measures of TIPN - heat thresold | At Baseline and after 6th and 12th taxane perfusion
  Quantitative sensory testing - heat thresold measurement at each hand and feet
Instrumental objective measures of TIPN - cold thresold | At Baseline and after 6th and 12th perfusions
  Quantitative sensory testing - cold thresold measure on each hand and feet
Instrumental objective measures of TIPN - vibration treshold | At Baseline and after 6th and 12th perfusion
  Quanitative sensory testing - vibration treshold
Instrumental objective meeasures of TIPN - electrochemical skin conductance (ESC) | At Baseline and after 6th and 12 perfusion
  Quantitative skin conductance testing - skin conductance measurements at each hand and feet

OTHER OUTCOMES:
Nail toxicity grading | At Baseline and before 4th and 12th perfusion
  Nail toxicity grading at each hand and foot : nail discoloration; nail riding; nail onycholysis - each graded as absent, mild, moderate or severe.

CONTACTS AND LOCATIONS:
Overall Officials: Janusz M Czernielewski, MD, PhD, Study Director — Tarian Pharma
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No